CLINICAL TRIAL: NCT06897072
Title: The Effect Of Yoga Applied In Childbirth Preparation Classes On Mode Of Delivery Preference, Bırth Satisfaction And Newborn Outcome: A Randomised Controlled Study
Brief Title: The Effect of Yoga on Labour and Neonatal Outcomes in Pregnant Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, SABRIYE UCAN YAMAC, Dr., Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GO 2024/838
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy Related
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Masking Description: They did not know if they were in the control and intervention group at the time of randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga (Experimental): It was planned to exclude those who did not accept to participate in the study, who were diagnosed with risky pregnancy, who were illiterate, who had systemic disease and mental problems requiring treatment, who had a gestational week less than 26-28, and who had communication and language problems. After the sampling is completed, the aims of the study will be explained to all pregnant women and they will be included in the study if they are satisfied. Participants in the experimental group will start the first pregnancy yoga session between the 26th and 28th weeks of pregnancy and attend the last session at the 37th week of pregnancy. They will practice yoga twice a week (each session lasting 75 minutes) in childbirth preparation classes
  Interventions: Behavioral: Yoga
- Control (No Intervention): The control group will receive the routine antenatal care that all pregnant women receive.

INTERVENTIONS:
Behavioral: Yoga — In the experimental group, yoga exercises were performed for 50 minutes with physical yoga movements (Vrksasana (tree pose), janusirsasana (head-knee pose), modifiedmarichyasana (great sage pose), baddhakonasana (connected angle pose), malasana (garland pose), sukhasana (meditation pose), ardhapadmasana (lotus sitting pose), gomukhasana (cow face pose), supta matyendrasana (spinal rotation pose on the back), bharmanasana (table pose), chakravasana (cat/cow pose), dandayamanabharmasana (balancing yoga pose), vajrasana (diamond pose), viraphadrasana 1-2 (warrior 1-2 pose). The class will include 15 minutes of meditation (deep relaxation with a focus on breath and self-awareness), breathing exercises in between and 10 minutes of relaxation.
  Arms: Yoga

SUMMARY:
The aim of this study was to determine the effect of yoga on mode of delivery preference, labour satisfaction and neonatal outcomes. This study was planned as a randomised controlled experimental study. The population of the study will consist of pregnant women who apply to the childbirth preparation classes of the institutions affiliated to the Bucak District Health Directorate, who meet the inclusion criteria and accept to participate in the study. The sample of the study; It will consist of pregnant women who apply for pregnancy follow-up to the birth preparation class determined between the dates of the study (15.01.2025 - 30.04.2025), who meet the criteria for admission to the study and who accept the study. The sample number was calculated by performing power analysis with the G power programme (19) and taking a study as a reference (20). According to the power analysis, the sample size was determined as 80 people (40 experimental, 40 control) to reach 95% power with an effect size of 0.8 and a 5% margin of error.

ELIGIBILITY:
Inclusion Criteria:

* being a woman
* who had a gestational week over than 26-28

Exclusion Criteria:

* who did not accept to participate in the study,
* who were diagnosed with risky pregnancy,
* who were illiterate,
* who had systemic disease and mental problems requiring treatment, who had a gestational week less than 26-28, and
* who had communication and language problems.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Birth Satisfaction Scale Revised Form (BSS-R) | up to 24 weeks
  In order to evaluate birth satisfaction, the Birth Satisfaction Scale Revised form (BSS-R) developed by a researcher was adapted into Turkish and a validity and reliability study was conducted. The BSS-R is a 5-point Likert-type scale. It is scored as strongly disagree '0 points', disagree '1 point', undecided '2 points', agree '3 points', strongly agree '4 points'. The lowest score of 0 and the highest score of 40 points can be obtained from the scale. In the scale, 6 statements are positive, 4 statements are negative and 4 items are reverse scored. The reverse scored items are items 2, 4, 7, 8. The higher the score obtained from the scale, the higher the woman's satisfaction with childbirth. In this study, the Cronbach's alpha reliability coefficients of the scale were 0.72 for BSS-R total, 0.78 for 'Quality of Care Services', 0.71 for 'Stress Experienced in Trauma', and 0.70 for 'Personal Characteristics of Women'.

SECONDARY OUTCOMES:
Scale of Pregnant Women's Preferences for Mode of Delivery | up to 24 weeks
  The scale was developed to determine the birth preferences of pregnant women based on the Health Belief Model and Planned Behaviour Model. The Turkish validity and reliability study was conducted. The scale is suitable for naturally pregnant women without systemic and psychiatric diseases. The scale consists of 18 items in total and three sub-dimensions (self-efficacy, normative beliefs, preferences). The scale form is 5-point Likert type. Each item in the scale is scored on the options of Strongly Disagree (1), Disagree (2), Undecided (3), Agree (4) and Strongly Agree (5).

CONTACTS AND LOCATIONS:
Locations (1):
- Burdur Mehmet Akif Ersoy University, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All authors contributed to the interpretation, writing, and approval of the final manuscript.

REFERENCES:
- [Result] Koyuncu SB, Bulbul M. The impact of yoga on fear of childbirth and childbirth self-efficacy among third trimester pregnants. Complement Ther Clin Pract. 2021 Aug;44:101438. doi: 10.1016/j.ctcp.2021.101438. Epub 2021 Jul 8. PMID 34252859
- [Result] Pais M, Pai MV, Kamath A, Bhat R, Bhat P, Joisa GH. A Randomized Controlled Trial on the Efficacy of Integrated Yoga on Pregnancy Outcome. Holist Nurs Pract. 2021 Sep-Oct 01;35(5):273-280. doi: 10.1097/HNP.0000000000000472. PMID 34407025
- [Result] Van der Riet P, Francis L, Rees A. Exploring the impacts of mindfulness and yoga upon childbirth outcomes and maternal health: an integrative review. Scand J Caring Sci. 2020 Sep;34(3):552-565. doi: 10.1111/scs.12762. Epub 2019 Dec 3. PMID 31797402